CLINICAL TRIAL: NCT04050072
Title: Patient-Reported Outcome Version of the Common Criteria for Adverse Events
Status: Active, not recruiting | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: PROSYM; 1R01CA238368-01A1 (NIH)
Record Dates: First submitted 2019-08-06; First posted 2019-08-08 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Survivorship; Cancer
Keywords: Adverse Events
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (3):
- Childhood Cancer Survivors (CCSS): i. PRO-CTCAE-SCC ii.Quality of life assessment
  Interventions: Other: Childhood Cancer Survivors (CCSS)
- St. Jude Life (SJLIFE): i. PRO-CTCAE-SCC ii. Quality of life assessment iii. Comprehensive medical evaluation, physical performance evaluation, and neurocognitive evaluation
  Interventions: Other: SJLIFE
- Community non-cancer control: i. PRO-CTCAE-SCC ii.Quality of life assessment
  Interventions: Other: Community non-cancer control

INTERVENTIONS:
Other: Childhood Cancer Survivors (CCSS) — To use the PRO-CTCAE-SCC (beta version) to identify symptomatic adverse event (AEs) that are prevalent and clinically meaningful in adult survivors of childhood cancer vs. non-cancer controls, and to create symptomatic AE items that are not included in the current PRO-CTCAE for adult survivors of childhood cancer.
  Other Names: Quality of life assessment; Late medical effects and health care utilization; Lifestyle assessment
  Groups: Childhood Cancer Survivors (CCSS)
Other: SJLIFE — To use the current PRO-CTCAE to conduct a symptom content creation process for the PRO-CTCAE-SCC by identifying clinically meaningful symptomatic AEs for adult survivors of childhood cancer, to create symptomatic AE items not included in the current PRO-CTCAE, and to perform comprehensive medical evaluation, physical performance evaluation, and neurocognitive evaluation to clinically validate the PRO-CTCAE-SCC.
  Other Names: Quality of life assessment; Comprehensive medical evaluation, physical performance evaluation, and neurocognitive evaluation
  Groups: St. Jude Life (SJLIFE)
Other: Community non-cancer control — To use the PRO-CTCAE-SCC (beta version) to identify symptomatic adverse event (AEs) that are prevalent and clinically meaningful in non-cancer controls vs. adult survivors of childhood cancer, and to create symptomatic AE items that are not included in the current PRO-CTCAE for adult survivors of childhood cancer.
  Other Names: Quality of life assessment; Late medical effects and health care utilization; Lifestyle assessment
  Groups: Community non-cancer control

SUMMARY:
Childhood cancer survivors are vulnerable to treatment-related late effects, including physical and psychosocial morbidities, subsequent malignancies, and premature death. Symptom assessment provides a unique insight into survivorship care since symptoms not only indicate the manifestation for the occurrence of chronic health conditions, but also impact quality of life and survival. The National Cancer Institute (NCI) has developed a Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) to assess symptomatic adverse events (AEs) for adult-onset cancer patients who are receiving cancer therapies. However, content-appropriate and clinically validated symptom assessment tools for adult survivors of childhood cancer are not available.

Primary Object 1: Establish content validity for the PRO-CTCAE-SCC

Primary Objective 1A: Conduct a symptom selection process through qualitative research to identify symptomatic AEs for adult survivors of childhood cancer

Primary Objective 1B: Create symptomatic AE items for adult survivors of childhood cancer based on the prevalence and clinical importance ratings on the items

Primary Objective 2: Validate the PRO-CTCAE-SCC using psychometric methods and objective clinical parameters

Primary Objective 2A: Test dimensionality for the PRO-CTCAE-SCC

Primary Objective 2B: Test clinical validity for the PRO-CTCAE-SCC

Primary Objective 2C: Test responsiveness to change for the PRO-CTCAE-SCC

Secondary Objective 1: Increase clinical usefulness of the PRO-CTCAE-SCC

Secondary Objective 2: Establish meaningful cut-points and minimally important differences (MIDs) on symptom burden scores for clinical decision-making

DETAILED DESCRIPTION:
We propose to adapt an existing symptomatic adverse event tool, the Patient-Reported Outcomes Common Terminology Criteria for Adverse Events (PRO-CTCAE), to be content appropriate and clinically meaningful for adult survivors of childhood cancer using two well-established childhood cancer survivor cohorts. Psychometric methodologies will be used to validate this tool by incorporating objective clinical anchors collected from medical evaluations. Our symptomatic AE tool has the potential to augment the Children Oncology Group Survivorship Care Guidelines by implementing risk-based symptom screening to track and anticipate adverse health events.

ELIGIBILITY:
Inclusion Criteria:

* > or equal to16 years of age at the time of enrollment
* > or equal to 5 years from initial diagnosis of pediatric cancer/malignancy (for CCSS and SJLIFE survivors only) and currently not receiving cancer therapies.

Exclusion Criteria:

* Have a known severe neurocognitive impairment, which requires proxies/parents to complete the survey
* Have < third grade reading level or are not able to communicate in English
* Unable to use and/or access internet or computer/tablet (for survey only)
* Unable to communicate and read in English

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All participants who meet eligibility criteria and consent to enrollment on the study.
Sampling Method: Probability Sample
Enrollment: 837 (Actual)
Dates: Start 2019-12-16 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
PRO-CTCAE-SCC | Years 1-5
  Conduct a symptom selection process through qualitative research to identify symptomatic AEs for adult survivors of childhood cancer, create symptomatic AE items for adult survivors of childhood cancer based on the prevalence and clinical importance ratings on the items, test dimensionality for the PRO-CTCAE-SCC, test clinical validity for the PRO-CTCAE-SCC and test responsiveness to change for the PRO-CTCAE-SCC.

SECONDARY OUTCOMES:
Core and Target Scales of the PRO-CTCAE-SCC | Years 4 and 5
  Develop tailored versions for survivors of different diagnoses exposed to different therapies and establish meaningful cut-points and minimally important differences (MIDs) on symptom burden scores for clinical decision-making.

CONTACTS AND LOCATIONS:
Overall Officials: I-Chang Huang, PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols